CLINICAL TRIAL: NCT06873516
Title: A Randomized, Double-Blind, Placebo Controlled, Dose-Ranging Study Evaluating the Efficacy and Safety of EVO756 in Adults With Moderate to Severe Chronic Spontaneous Urticaria
Brief Title: Phase 2b Study of EVO756 in Adults With Moderate to Severe Chronic Spontaneous Urticaria (CSU)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Evommune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVO756-CSU001
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: chronic spontaneous urticaria; CSU; chronic hives; hives; idiopathic urticaria; urticaria
MeSH Terms: conditions — Chronic Urticaria; Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose 1 (Experimental): Orally administered EVO756, dose 1
  Interventions: Drug: EVO756
- Dose 2 (Experimental): Orally administered EVO756, dose 2
  Interventions: Drug: EVO756
- Dose 3 (Experimental): Orally administered EVO756, dose 3
  Interventions: Drug: EVO756
- Placebo control (Placebo Comparator): Orally administered placebo control
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: EVO756 — Dose 1
  Arms: Dose 1
Drug: EVO756 — Dose 2
  Arms: Dose 2
Drug: EVO756 — Dose 3
  Arms: Dose 3
Drug: Placebo control — Placebo control
  Arms: Placebo control

SUMMARY:
This study will evaluate the efficacy and safety of different doses of EVO756 in adults with moderate to severe chronic spontaneous urticaria (CSU).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed CSU diagnosis for at least 3 months with an inadequate response to H1-antihistamines.
* Subjects who are taking H1-antihistamines must be on a stable regimen 4 weeks prior to Day 1 and while on study.
* Urticaria Activity Score (UAS7) equal to or greater than 16 at Day 1. UAS entries must be completed for a minimum of 4 out of the 7 days prior to Day 1.

Exclusion Criteria:

* Any clinically significant abnormality in laboratory evaluations, physical examinations, vital signs, or ECG at Screening, according to the Investigator's discretion.
* Use of certain medications.
* History of diseases with urticaria or angioedema symptoms, other than CSU and symptomatic dermographism.
* Significant medical history other than CSU, or any other condition which might interfere with the evaluation of CSU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in UAS7 | Week 12

SECONDARY OUTCOMES:
Percent change from baseline in UAS7 | Week 12
Mean and percent change from baseline in UAS7 | Weeks 1, 2, 4, 8
Mean and percent change from baseline in ISS7 | Weeks 1, 2, 4, 8, 12
Mean and percent change from baseline in HSS7 | Weeks 1, 2, 4, 8, 12
Mean and percent change from baseline in AAS7 | Weeks 1, 2, 4, 8, 12
Proportion of subjects achieving UAS7 ≤ 6 | Weeks 1, 2, 4, 8, 12
Proportion of subjects achieving UAS7 = 0 | Weeks 1, 2, 4, 8, 12

CONTACTS AND LOCATIONS:
Locations (53):
- United States (41):
  - Cahaba Dermatology Skin Health Center, Birmingham, Alabama
  - Velocity Clinical Research, Mobile, Mobile, Alabama
  - Center for Dermatology Clinical Research, Fremont, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Northridge Clinical Trials, Northridge, California
  - NorthBay Clinical Research, Santa Rosa, California
  - Integrated Research of Inland, Upland, California
  - FOMAT Medical Research, Ventura, California
  - AMR Fort Myers, Fort Myers, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - Sneeze, Wheeze & Itch Associates LLC, Normal, Illinois
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - The Iowa Clinic, West Des Moines, Iowa
  - Hutchinson Clinic, Hutchinson, Kansas
  - Bluegrass Allergy Care, Lexington, Kentucky
  - Delricht Research Louisville, Louisville, Kentucky
  - Delricht Research Louisiana, Baton Rouge, Louisiana
  - Velocity Clinical Research, Lafayette, Lafayette, Louisiana
  - Delricht Research, New Orleans, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Boston Specialists, Boston, Massachusetts
  - MI Skin Innovations, Northville, Michigan
  - DelRicht Research - Town Center Dermatology, Wildwood, Missouri
  - Vitality Clinical Trials, Woodbury, New York
  - Allergy Partners Clinical Research, Asheville, North Carolina
  - Delricht Research - Priority Care, Charlotte, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Optima Research Boardman, Boardman, Ohio
  - DOCS Dermatology Research, Canal Winchester, Ohio
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - AMR Myrtle Beach, Myrtle Beach, South Carolina
  - National Allergy and Asthma Research, North Charleston, South Carolina
  - Delricht Research Smyrna, Smyrna, Tennessee
  - Austin Regional Clinic ARC Clinical Research, Austin, Texas
  - Studies in Dermatology, Cypress, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Delricht Research - Lockhard Matter Dermatology, Prosper, Texas
  - AMR Utah, Layton, Utah
  - Seattle Clinical Research Center, Seattle, Washington
  - Allergy, Asthma, and Sinus Center, Greenfield, Wisconsin
- Canada (5):
  - Dandelion Allergy Centre, Mississauga, Ontario
  - Allergy Research Canada, Niagara Falls, Ontario
  - Red Maple Trials, Ottawa, Ontario
  - Centre de Recherche Saint-Louis - Montréal, Montreal, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec
- Japan (7):
  - Dermatology and Ophthalmology Kume Clinic, Sakai, Osaka
  - Yoshikawa Skin Clinic, Takatsuki, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - Mita Dermatology, Minato-Ku, Tokyo
  - ThinkPark Dermatology Clinic, Shinagawa-Ku, Tokyo
  - Medical Corporation Jitai-kai Tachikawa Dermatology Clinic, Tachikawa, Tokyo
  - Ikebukuro Nishiguchi Fukurou Dermatology, Toshima-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No